CLINICAL TRIAL: NCT04869319
Title: Electronic Triggers: Messaging After A1C EHR Alert
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: QI-A1C
Record Dates: First submitted 2021-03-18; First posted 2021-05-03 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Hemoglobins; Diagnostic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MyChart message: MyChart message subjects with high A1C blood tests to help manage their diabetes and prevent some of the complications caused by high sugars. The message recommends that they schedule a visit with their doctor who can recheck the blood test and help get their diabetes under control.
  Interventions: Behavioral: MyChart message
- No MyChart message: No message

INTERVENTIONS:
Behavioral: MyChart message — Message subjects through MyChart to follow-up with their provider to schedule a follow up HbA1C test.
  Groups: MyChart message

SUMMARY:
Studying subjects with HbA1C tests >10 and no follow-up test within 6 months and appointments scheduled in the next 60 days from data run date. Subjects who receive intervention message may be more likely to follow up with their provider to schedule a follow up HbA1C test.

ELIGIBILITY:
Inclusion Criteria:

* MyChart active patients with HbA1C tests >10 and no follow-up test within 6 months and no appointments scheduled in the next 60 days from data run date

Exclusion Criteria:

* Patients with a scheduled appointment within 60 days from time algorithm is run; hospital encounters; non English or Spanish patients as indicated by primary language in Epic

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MyChart active patients with HbA1C tests >10 and no follow-up test within 6 months and no appointments scheduled in the next 60 days from data run date
Sampling Method: Probability Sample
Enrollment: 2403 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Rate of follow up A1C within 9 months after original A1C (allowing 3 months after email is sent) | 2 years
  This outcome measures the rate at which participants complete an A1C test within 3 months of the message intervention being sent and 9 months of their original test.

CONTACTS AND LOCATIONS:
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No